CLINICAL TRIAL: NCT07269509
Title: Evaluation of the Efficacy and Safety of an Intensified Strategy of Intratonsillar Immunotherapy (ITIT) for Allergic Rhinitis: A Multicenter, Randomized, Double-blind, Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WDRY2025-K209(X01)
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinitis; Intratonsillar; Allergen immunotherapy; Standardized dust mite allergen extracts
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Inject mite allergen solution into the tonsil at the 0th, 1st, 2nd, 6th, 12th, 18th and 24th months.
  Interventions: Procedure: Strengthen Intratonsillar Immunotherapy (ITIT)
- control group (Placebo Comparator): Inject the mite allergen solution into the tonsil at months 0, 1, 2, 12, and 24, and administer the placebo at months 6 and 18.
  Interventions: Procedure: Basic Intratonsillar Immunotherapy (ITIT)

INTERVENTIONS:
Procedure: Basic Intratonsillar Immunotherapy (ITIT) — During injection, the operator needs to gently shake the injection bottle about 20 times, the drug must be mixed to ensure the consistency of allergen concentration, and carefully check the patient's name and concentration on the bottle. Allergy extracts should not be injected intravenously, so the syringe will be aspirated to avoid inadvertent intravascular injection. Before each injection, after inserting the needle into the selected tonsil, before injecting the dose, the investigator will slightly pull the plunger of the syringe. If blood returns from the syringe, the syringe, and its contents will be discarded. The other tonsil will be selected and a new syringe will be prepared.
  Inject the mite allergen solution into the tonsil at months 0, 1, 2, 12, and 24, and administer the placebo at months 6 and 18.
  Arms: control group
Procedure: Strengthen Intratonsillar Immunotherapy (ITIT) — During injection, the operator needs to gently shake the injection bottle about 20 times, the drug must be mixed to ensure the consistency of allergen concentration, and carefully check the patient's name and concentration on the bottle. Allergy extracts should not be injected intravenously, so the syringe will be aspirated to avoid inadvertent intravascular injection. Before each injection, after inserting the needle into the selected tonsil, before injecting the dose, the investigator will slightly pull the plunger of the syringe. If blood returns from the syringe, the syringe, and its contents will be discarded. The other tonsil will be selected and a new syringe will be prepared.
  Inject mite allergen solution into the tonsil at the 0th, 1st, 2nd, 6th, 12th, 18th and 24th months.
  Arms: experimental group

SUMMARY:
This is a multicenter, randomized, double-blind, controlled trial to evaluate the efficacy and safety of an enhanced strategy of allergen-specific immunotherapy (ITIT) in the treatment of allergic rhinitis. By recording the changes in CSMS from baseline to post-treatment in the subjects and the incidence of adverse reactions after treatment, the differences in efficacy and safety between the patients who received the basic three doses and those who received booster injections were compared. Furthermore, the impact of different booster strategies on long-term efficacy was compared to optimize the injection strategy. At the same time, the influence of different administration procedures on the immune response was evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signing of the informed consent form
2. Commitment to abide by the research procedures and cooperate throughout the implementation of the research
3. Diagnosis conforms to the ARIA guidelines. The basis for the diagnosis is as follows: a. Symptoms: Paroxysmal sneezing, clear nasal discharge, nasal itching, and nasal congestion occur for 2 or more times, with symptoms persisting or accumulating for more than 1 hour each day, accompanied by tearing, eye itching, and eye redness and other ocular symptoms; b. Signs: Commonly, the nasal mucosa is pale and edematous, and nasal watery secretions are present; c. Allergen testing: Positive results for dust mite allergens SPT and/or serum-specific IgE, or positive nasal challenge test, requiring Der p and Der f to be positive (SPT results of ++ or higher, serum sIgE ≥ 2 grades), and other allergens in the allergen test to be negative
4. History of allergic rhinitis caused by atopic dust mite allergens
5. Infertile women must ensure they do not become pregnant during the treatment period
6. Age must be between 5 and 60 years old

Exclusion Criteria:

1. Allergic to the excipients of Arrogel (aluminum hydroxide) or the rescue medication epinephrine
2. Suffering from respiratory system diseases other than stable asthma
3. Pulmonary dysfunction (NYHA grade II or above, or FeV1 < 70%) or having irreversible pathological changes in the reactive organs such as emphysema or bronchiectasis
4. Severe acute or chronic diseases (including malignant diseases), inflammation and fever
5. Multiple sclerosis
6. Immune system diseases (autoimmune diseases, immune diseases caused by antigen-antibody complexes, immune deficiencies, etc.)
7. Active pulmonary tuberculosis
8. Severe mental disorders
9. Obvious cardiac dysfunction
10. Patients who have received immunotherapy within the last 1 years (subcutaneous injection or sublingual administration of allergen-specific immunotherapy, etc.)
11. Patients who used experimental drugs or participated in other clinical studies within 30 days before treatment
12. Patients who received IgE monoclonal antibody (mAb) treatment in the past 4 months
13. Patients taking beta-blockers
14. Patients who have insufficient understanding of the trial
15. Patients whose age is not between 5 years old and 65 years old
16. Patients who are pregnant or breastfeeding during the study period, or have plans to get pregnant
17. Patients who cannot undergo tonsil injection due to acute or chronic tonsillitis, small tonsils, previous tonsillectomy, overly sensitive pharyngeal reflex and inability to cooperate with treatment
18. Patients with aphthous stomatitis

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
CSMS | Before treatment (baseline) and at 1, 2, 3, 6, 12, 24, and 36 months after treatment.
  combined symptom and medication score
adverse event | 30 minutes after each treatment (at the 0th, 1st, 2nd, 6th, 12th, 18th and 24th months).
  Observe adverse events and classify them according to the World Allergy Organization (WAO) subcutaneous immunotherapy reaction classification system.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | Before treatment (baseline) and at 1, 2, 3, 6, 12, 24, and 36 months after treatment.
  Pain perception of allergy symptoms during treatment will be evaluated using a scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates maximum pain.
Absolute Value and Percentage of Blood Leukocytes | Before treatment (baseline) and at 6, 12, 24, and 36 months after treatment.
Concentration of Key Serum Cytokines | Before treatment (baseline) and at 6, 12, 24, and 36 months after treatment.
Concentration of Serum Immune Globulins | Before treatment (baseline) and at 6, 12, 24, and 36 months after treatment.
Proportion of T Cell Differentiation | Before treatment (baseline) and at 6, 12, 24, and 36 months after treatment.
ARCT | At 1, 2, 3, 6, 12, 24, and 36 months after treatment.
  The Allergic Rhinitis Control Test Questionnaire
miniRQLQ | Before treatment (baseline) and at 1, 2, 3, 6, 12, 24, and 36 months after treatment.
  mini Rhinoconjunctivitis Quality of Life Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
Two years after the completion of the trial, data will be published on the EDC (http://edc.eplat.com.cn/).
Supporting Information: Study Protocol, CSR
Time Frame: Two years after the completion of the trial
Access Criteria: Upon approval of the request, access to the de-identified individual patient-level data will be provided. Before accessing the requested information, a data sharing agreement (a non-negotiable contract for data visitors) must be signed.
URL: http://edc.eplat.com.cn/

REFERENCES:
- [Background] Gu T, Zhang W, Tan L, Xiang R, Liu P, Huang J, Deng Q, Deng Y, Tao Z, Chen S, Xu Y. Intratonsillar Immunotherapy: A Convenient and Effective Alternative to Subcutaneous Immunotherapy for Allergic Rhinitis. Research (Wash D C). 2025 Jan 16;8:0573. doi: 10.34133/research.0573. eCollection 2025. PMID 39822282
- See also: Related Info — https://www.medicalresearch.org.cn/